CLINICAL TRIAL: NCT03179332
Title: A Euglycaemic Clamp Trial to Evaluate the Pharmacokinetic and Pharmacodynamic Properties of a Bolus Dose of BioChaperone® Insulin Lispro, Fiasp® and NovoRapid® by an Insulin Pump
Brief Title: A Trial to Evaluate the Pharmacokinetic and Pharmacodynamic Properties of BioChaperone® Insulin Lispro, Fiasp® and NovoRapid® Delivered by an Insulin Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT032-ADO02
Record Dates: First submitted 2017-05-04; First posted 2017-06-07 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BioChaperone® insulin lispro (Experimental): Single subcutaneous administration of BioChaperone® insulin lispro
  Interventions: Drug: BioChaperone® insulin lispro
- Fiasp® (Active Comparator): Single subcutaneous administration of Fiasp® (insulin aspart)
  Interventions: Drug: Fiasp®
- Novorapid® (Active Comparator): Single subcutaneous administration of Novorapid® (insulin aspart)
  Interventions: Drug: Novorapid®

INTERVENTIONS:
Drug: BioChaperone® insulin lispro — Single subcutaneous administration of a bolus of 0.15 U/kg body with a pump
  Arms: BioChaperone® insulin lispro
Drug: Fiasp® — Single subcutaneous administration of a bolus of 0.15 U/kg body with a pump
  Arms: Fiasp®
Drug: Novorapid® — Single subcutaneous administration of a bolus of 0.15 U/kg body with a pump
  Arms: Novorapid®

SUMMARY:
This is a single-centre, randomised, double-blind, three-period, complete cross-over trial comparing the pharmacokinetic and the pharmacodynamic properties of BioChaperone® insulin lispro and the two active comparators Fiasp® and Novorapid® when given as a bolus on top of basal delivery with an insulin pump in subjects with type 1 diabetes mellitus. Each subject will be randomly assigned to a treatment sequence consisting of 3 dosing visits during which the subject will receive the investigational products. In a euglycaemic clamp setting, subjects will be given a bolus dose of 0.15 U/kg body weight.

Throughout the glucose clamp procedure, blood glucose will be stabilised at a target level of 100 mg/dL by means of an intravenous infusion of glucose. Blood samples for pharmacokinetic assessment will be drawn at specified timepoints and glucose infusion rates and blood glucose concentrations will be recorded for pharmacodynamic assessment during the 10-hour clamp procedure after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus for more than 12 months.
* BMI between 18.5 and 28.5 kg/m².
* HbA1C level <=9.0%.
* Insulin treated for at least 12 months with total insulin dose <1.2U/kg/day.

Exclusion Criteria:

* Type 2 Diabetes Mellitus.
* History of multiple and/or severe allergies to drugs or foods.
* Any history or presence of clinically relevant cardiovascular, pulmonary, respiratory, gastrointestinal, hepatic, renal, metabolic, endocrinological (with the exception of conditions associated with diabetes mellitus), haematological, dermatological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness as judged by the Investigator.
* More than one episode of severe hypoglycaemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Proliferative retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy.
* Females of childbearing potential, who are pregnant, breast-feeding or intend to become pregnant or are not using highly effective contraceptive methods.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
AUCGIR(0-60min) | 60 minutes
  Baseline corrected area under the glucose infusion rate curve from 0 to 60 minutes after bolus administration

SECONDARY OUTCOMES:
AUCins(0-30min) | 30 minutes
  Baseline corrected area under the insulin concentration time curve from 0 to 30 minutes after bolus administration
AUCins(0-60min) | 60 minutes
  Baseline corrected area under the insulin concentration time curve from 0 to 60 minutes after bolus administration
AUCins(0-600min) | 600 minutes
  Baseline corrected area under the insulin concentration time curve from 0 to 600 minutes after bolus administration
Cmax insulin | 10 hours
  Maximum observed baseline corrected insulin concentration
Tmax insulin | 10 hours
  Time from bolus administration to baseline corrected Cmax
TmaxGIR | 10 hours
  Time from bolus administration to maximum baseline corrected glucose infusion rate
GIRmax | 10 hours
  Maximum baseline corrected glucose infusion rate
Adverse Events | up to 8 weeks
  Number of Adverse Events in each arm
Clinical safety laboratory | up to 8 weeks
  Haematology, biochemistry and urinalysis: changes and findings from Baseline in clinical safety laboratory parameters during the trial duration, from screening, and at follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No